CLINICAL TRIAL: NCT00150150
Title: Ultrasound Guided Interstitial Laser Photocoagulation on Benign Thyroid Nodules
Brief Title: Laser Therapy of Benign Thyroid Nodules
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 017
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Benign Solitary Solid; Cystic Thyroid Nodules
Keywords: Interventional ultrasound; interstitial laser theraphy; tumor ablation; nodule reduction; adverse effects; patient satesfaction

INTERVENTIONS:
Procedure: Interstitial laser photocoagulation

SUMMARY:
Nodular goitre is common in the general population and less than 5% of the patients who undergo surgery for solitary thyroid nodules have cancer, in absence of clinical suspicion. Nodules left untreated seem to have a slight growth potential in borderline iodine-deficient areas. Interstitial laser photo-coagulation (ILP) is a procedure for local hyperthermia and photocoagulation, allowing minimally invasive treatment of benign tumors, including thyroid nodules. The aim of these studies are to evaluate if ILP will be useful in reducing the volume of the benign thyroid nodule and thyroid function will be unaffected in euthyroid patients, and normalized in pretoxic- and toxic thyroid nodules. The investigations are listed below:

1. Randomized study of interstitial laser photocoagulation for benign solitary cold thyroid nodules - one versus two or three treatments
2. Randomized study of interstitial laser photocoagulation for benign solitary autonomous thyroid nodules - 131I versus laser ablation
3. Interstitial laser photocoagulation for benign thyroid cystadenomas. - a feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a solitary solid thyroid nodule confirmed by ultrasonography
* Patients with a solitary cystadenoma (cystic part more than 2 mL) confirmed by ultrasonography
* Patients with an autonomous functioning thyroid nodule.

Exclusion Criteria:

* No family history of thyroid cancer
* Prior radiation towards the neck
* Fine needle biopsy without valid diagnostic criteria for benign thyroid disease
* Nodules larger than 4 cm (largest diameter)
* Suspicion of malignancy
* Increased serum calcitonin
* Pregnancy or lactation
* Alcohol, medicine or drug abuse
* No safe contraception
* Physical or psychic condition that hinders corporation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2001-01; Study Completion 2006-03

PRIMARY OUTCOMES:
To evaluate the efficacy and feasibility repeated ILP treatments in a prospective randomised study where the nodule and thyroid volume are measured 1, 3, 6 and 12 months after the ILP.
In the study of patients with a cystadenoma the measures will be done like wise, but also the recurrence of the cystic part will be measured.
Patients with an autonomous functioning nodule measurements of thyroid function are performed 1,2, 3, 6, 9 and 12 months after the ILP or 131I therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Døssing, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark